CLINICAL TRIAL: NCT03245333
Title: Phase Ⅲ Clinical Study of Recombinant Human Growth Hormone Injection (JINTOPIN AQ) for Short Children With Small for Gestational Age(SGA)
Brief Title: A Study of Recombinant Human Growth Hormone Injection for Short Children With Small for Small for Gestational Age(SGA)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Tongji Hospital (Other); Beijing Children's Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Shanghai Children's Hospital (Other); The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GenSci 030 CT-III
Record Dates: First submitted 2017-07-18; First posted 2017-08-10 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-07

CONDITIONS: Small for Gestational Age Infant
MeSH Terms: interventions — Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Stage 1-experimental group (Experimental): JINTOPIN AQ 0.2IU/kg/d（0.46mg/kg /wk）, for 52 weeks.
  Interventions: Drug: Recombinant Human Growth Hormone Injection
- Stage 1-negative control (Other): observed only for 52 weeks.
  Interventions: Drug: Recombinant Human Growth Hormone Injection
- Stage 2-experimental group (Experimental): After completing the stage 1, experimental groups is administrated the appropriate dose of JINTOPIN AQ, the highest dose should be no more than 0.2IU/kg/d, from the 53rd week to the final height.
  Interventions: Drug: Recombinant Human Growth Hormone Injection
- Stage 2-negative control (Other): After completing the stage 1, negative control groups is administrated the appropriate dose of JINTOPIN AQ, the highest dose should be no more than 0.2IU/kg/d, from the 53rd week to the final height.
  Interventions: Drug: Recombinant Human Growth Hormone Injection

INTERVENTIONS:
Drug: Recombinant Human Growth Hormone Injection — Stage 1：JINTOPIN AQ 0.2IU/kg/d（0.46mg/kg /wk）for 52 weeks.
  Other Names: rhGH Injection
Drug: Recombinant Human Growth Hormone Injection — Stage 2: After completing phase 1, patients are administrated the appropriate dose of JINTOPIN AQ, the highest dose should be no more than 0.2IU/kg/d, from the 53rd weeks to the final height.
  Other Names: rhGH Injection

SUMMARY:
According to the results of the phase II study, choose the best dose of JINTOPIN AQ for short SGA children, further to evaluate the efficacy and safety of the treatment of short SGA children.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of full-term small for gestational age, SGA.
* Chronological age between 2-6.5 years in girls and 2-7.5 years in boys. Both genders.
* Prepubertal stage (Tanner I).
* Height was lower than the mean -2SD of the values of normal children of the same age and gender when participating in the study.
* A GH peak concentration >10µg/L in a provocative test within a year before participating in the study.
* Bone age<Chronological age+1.
* Normal glucose regulation：Fasting blood-glucose < 5.6mmol/L, and 2 hours postprandial blood-glucose < 7.8mmol/L.
* Gestational age was 37 to 42 weeks.
* The subjects and their guardians signed informed consent.

Exclusion Criteria:

* Subjects with Liver and renal insufficiency (ALT > 1.5 times of upper limit of normal value, Cr> upper limit of normal value).
* Patients are positive for antibodies to hepatitis B core (HBc), hepatitis B surface antigen (HBsAg) or hepatitis B e antigen (HBeAg).
* Known Highly allergic constitution or allergic to the test drug.
* Subjects with diabetes, severe cardiopulmonary and pulmonary disease, and hematological diseases, malignant tumors, or systemic infection, immunocompromised patients and patients with psychosis.
* Subjects with other growth disorders, such as Turner syndrome, constitutional delay of growth and puberty, and Laron syndrome and growth hormone receptor deficiency.
* Subjects who have received the treatment of GH.
* Subjects took part in other clinical trial study within 3 months.
* Children who have treated with other hormone (such as gonadal hormone and glucocorticoids etc, continuous administration of more than a month) and that may affect growth hormone secretion or action including oxygen male dragon, growth hormone releasing hormone, etc. within 3 months.
* Other conditions which in the opinion of the investigator preclude enrollment into the study.

Ages: 24 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-12 (Actual); Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change of height standard deviation score for chronological age (△Ht SDSCA) | 52 weeks
  △Ht SDS= Ht SDSafter treatment - Ht SDSbaseline Ht SDSCA = (height - reference mean for CA) / reference SD for CA (refers to the height value at particular timepoint )

SECONDARY OUTCOMES:
Height（Ht）at the end of treatment | Stage 1：52 weeks
Height（Ht）at the end of treatment | Stage 2：Every 52 weeks, up to 3 years
Annualized height velocity (HV) | Stage 1：52 weeks
Annualized height velocity (HV) | Stage 2：Every 52 weeks, up to 3 years
Bone age maturation | Stage 1：52 weeks
Bone age maturation | Stage 2：Every 52 weeks, up to 3 years
Mole ratio of IGF-1 and IGFBP-3 | Stage 1：52 weeks
Mole ratio of IGF-1 and IGFBP-3 | Stage 2：Every 52 weeks, up to 3 years
IGF-1 standard deviation score (SDS) | Stage 1：52 weeks
IGF-1 standard deviation score (SDS) | Stage 2：Every 52 weeks, up to 3 years

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Tongji Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - The first affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - The Children's Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Beijing Children's Hospital, Capital Medical University, Beijing
  - Shanghai Children's Hospital, Shanghai